CLINICAL TRIAL: NCT06172764
Title: Effect of Vitamin D Supplementation on Salivary Biomarkers; Certain Proteins and Cariogenic Oral Microbiome for Medical Management of Dental Caries: A Randomized Controlled Trial
Brief Title: A Randomized Controlled Trial of Vitamin D Supplementation on Salivary Biomarkers and Cariogenic Oral Microbiome
Acronym: Incipient
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Collaborators: University of Karachi (Other)
Responsible Party: Principal Investigator, Saba Arshad, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SArshad
Record Dates: First submitted 2023-12-12; First posted 2023-12-15 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Dental Caries; White Spot Lesion; Initial Caries; Incipient Enamel Caries
Keywords: Dental Caries; White Spot Lesion; Initial Caries; Incipient Enamel Caries
MeSH Terms: conditions — Dental Caries | interventions — Behavior Therapy; Fluoride Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): vitamin D Deficient group having initial caries
  Interventions: Dietary Supplement: Vitamin D supplements along with behavioral modification
- Group B (Active Comparator): vitamin D deficient group having initial caries
  Interventions: Combination Product: Topical fluoride application and Vitamin D supplements along with behavioral modification
- Group C (Placebo Comparator): vitamin D sufficient group having initial caries
  Interventions: Procedure: Topical fluoride application along with behavioral modification

INTERVENTIONS:
Dietary Supplement: Vitamin D supplements along with behavioral modification — Vitamin D soft gel capsules of 50,000 IU/week for two months followed by a maintenance dosage of 5000 IU/day for one month.
  Behavior modification for dental caries with standard instructions of brushing teeth twice daily with regular fluoridated toothpaste and diet counseling.
  Arms: Group A
Combination Product: Topical fluoride application and Vitamin D supplements along with behavioral modification — Professional topical 5% sodium fluoride gel application for 5 minutes on the teeth having ICL.
  Behavior modification for dental caries with standard instructions of brushing teeth twice daily with regular fluoridated toothpaste and diet counseling.
  Vitamin D soft gel capsules of 50,000 IU/week for two months followed by a maintenance dosage of 5000 IU/day for one month.
  Behavior modification for dental caries with standard instructions of brushing teeth twice daily with regular fluoridated toothpaste and diet counseling.
  Arms: Group B
Procedure: Topical fluoride application along with behavioral modification — Professional topical 5% sodium fluoride gel application for 5 minutes on the teeth having ICL.
  Behavior modification for dental caries with standard instructions of brushing teeth twice daily with regular fluoridated toothpaste and diet counseling.
  Behavior modification for dental caries with standard instructions of brushing teeth twice daily with regular fluoridated toothpaste and diet counseling.
  Arms: Group C

SUMMARY:
The goal of this clinical trial is to compare the treatment effect of vitamin D supplementation and topical fluorides in the population having vitamin D deficiency and Initial Carious Lesions (ICL) on the progression of ICL in teeth. This study aims to observe the changes in the International Caries Detection and Assessment System (ICDAS) scores, the concentration of salivary proteins, and cariogenic microbes, six months after the interventions.

* Group A will get vitamin D supplements and oral hygiene instructions (OHI).
* Group B will get vitamin D supplements, topical fluorides, and OHI.
* Group C (Control), the vitamin D sufficient group will get topical fluorides and OHI.

DETAILED DESCRIPTION:
The study investigator will conduct a multi-centered randomized clinical trial in the outpatient department of Operative Dentistry, in three units of Dow University of Health Sciences (DUHS), with parallel treatment assignment to an experimental, active comparator, and control groups. The investigator will recruit study participants aged 12 to 45 at moderate risk of dental caries, specifically those with vitamin D deficiency. Additionally, participants must have at least two clinically diagnosed teeth with initial carious lesions (ICL). Each participant will be enrolled for six months in this trial.

The investigator will obtain data on vitamin D deficiency from Dow Diagnostic Laboratory. Dental caries risk will be assessed using a caries risk assessment (CRA) form, while ICL will be evaluated through the International Caries Detection and Assessment System (ICDAS) scores. The investigator will collect the samples of participants' saliva to analyze salivary proteins using the enzyme-linked immunosorbent assay (ELISA), and cariogenic microbes through polymerase chain reaction (PCR).

Participants will be assigned to one of three groups randomly:

* Group A participants will be vitamin D deficient with caries, receiving vitamin D supplements and Oral hygiene instructions (OHI).
* Group B participants will be vitamin D deficient with caries, receiving vitamin D supplements, topical fluorides, and OHI.
* Group C participants will be vitamin D sufficient to be considered as controls for comparison, receiving fluoride application and OHI.

The investigator will assess study outcomes by observing changes in ICDAS scores, salivary protein concentrations, and count of cariogenic bacterial species (Streptococcal mutans and Lactobacilli).

ELIGIBILITY:
Inclusion Criteria:

* Patients of all genders and ages ranging from 12-50 years, having at least two teeth with clinically diagnosed Initial Carious Lesions at Moderate Risk of Dental Caries, after written informed consent.
* Patients having vitamin D deficiency.

Exclusion Criteria:

* Patients who have heavy calculus, gingivitis, or periodontitis.
* Patients using desensitizing toothpaste or mouthwash up to six weeks before the study.
* Patients who have severe intestine or kidney disease, malabsorption syndrome, or any other conditions affecting vitamin D metabolism.
* Patients on antibiotics or probiotics therapy for the last month
* Pregnant females.
* Patients with poor oral hygiene and with excessive dietary exposure to acids and carbohydrates.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ICDAS scores of initial caries or white spot lesions | 6 months
  Change in ICDAS scores of initial caries or white spot lesions
Number of growth forming units of microbial strains | 6 months
  Change in number of growth forming units of microbial strains
Genetic expression of target genes of S. Mutans and L. Rhamnosus | 6 months
  Presence or absence of genetic expression of target genes of S. Mutans and L. Rhamnosus

SECONDARY OUTCOMES:
Serum Vitamin D levels | 6 months
  Change in Serum Vitamin D levels
Salivary protein concentration | 6 months
  Change in salivary protein concentration

CONTACTS AND LOCATIONS:
Overall Officials: Dr Saba Arshad, Principal Investigator — DUHS
Locations (1):
- Dr Saba Arshad, Karachi, Sindh, Pakistan